CLINICAL TRIAL: NCT02382367
Title: Prevalence of Alpha-1 Antitrypsin Dysfunction in Pulmonary Emphysema
Acronym: DysA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013.835
Record Dates: First submitted 2014-12-04; First posted 2015-03-06 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Pulmonary Emphysema
MeSH Terms: conditions — Pulmonary Emphysema | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pulmonary emphysema (Experimental): Blood tests (Alpha-1 antitrypsin protein measurement, elastase-inhibitory capacity of plasma measurement, phenotypic and genotypic studies)
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Blood tests (Alpha-1 antitrypsin protein measurement, elastase-inhibitory capacity of plasma measurement, phenotypic and genotypic studies)

SUMMARY:
The main objective of this trial is to evaluate the prevalence of alpha-1 antitrypsin quantitative and functional deficiency in an adult French population presenting with pulmonary emphysema. Phenotypic and genotypic studies will be carried whenever quantitative and/or functional deficiency will be displayed.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary emphysema highlighted by computed tomography
* Ratio Forced Expiratory Volume in 1 second (FEV1) / Vital Capacity (VC) < 70% measured by lung function test

Exclusion Criteria:

* Hepatic transplant
* Patient under legal protection
* Patient not benefiting from the French Health Insurance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of patient with alpha-1 antitrypsin dysfunction | Samples for evaluation of alpha-1 antitrypsin dysfunction will be performed the day of the patient enrollment
  Alpha-1 antitrypsin protein will be measured either on serum or plasma by standardized immunoassay. The elastase-inhibitory capacity of plasma will be evaluated by a functional test. The anti-elastase dysfunction of alpha-1 antitrypsin will be evaluated using both measurements.

SECONDARY OUTCOMES:
Determination of alpha-1 antitrypsin protein phenotype | Samples for phenotype analysis will be performed the day of the patient enrollment
  The determination of the alpha-1 antitrypsin protein phenotype may highlight genotype variants. The different known phenotypes are: Pi MM, Pi Z; Pi S, Pi SS, Pi SZ, Pi ZZ.
Molecular genotyping of gene coding alpha-1 antitrypsin | Samples for molecular genotyping will be performed the day of the patient enrollment
  For those patients who presented with either a functional or a quantitative dysfunction, we will look for genetic mutations in the gene coding the alpha-1 antitrypsin allowing the identification of specific genotype such as MM, MZ, MS, SS and SZ

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Louis Pradel - service de pneumologie, Bron, France